CLINICAL TRIAL: NCT01061242
Title: Post-ICU Neurocognitive Performance and Sleep Quality Ratings Following Exposure to a Medical ICU Sleep Quality Improvement Project
Brief Title: Intensive Care Unit (ICU) Sleep Quality and Neurocognitive Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Dale M. Needham, MD, PhD, Johns Hopkins University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NA_00033951
Record Dates: First submitted 2010-02-02; First posted 2010-02-03 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2009-12

CONDITIONS: Neurobehavioral Manifestations; Sleep Deprivation; Dyssomnias
Keywords: Neurocognitive function; Sleep quality; Critical care; Quality Assurance, health care
MeSH Terms: conditions — Neurobehavioral Manifestations; Sleep Deprivation; Dyssomnias; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Baseline (No Intervention): Post-Intensive Care Unit (ICU) neurocognitive testing and sleep survey performed on patients exposed to ad-lib Medical ICU environment.
- Sleep Promotion Group (Experimental): Post-ICU neurocognitive testing and sleep survey performed on patients exposed to interventions in the pre-existing MICU sleep quality improvement project.
  Interventions: Behavioral: Sleep promoting interventions

INTERVENTIONS:
Behavioral: Sleep promoting interventions — MICU staff will implement multi-faceted, staged sleep promoting interventions as part of a pre-existing sleep quality improvement project.
  Arms: Sleep Promotion Group

SUMMARY:
The purpose of this study is to understand patients' neurocognitive performance shortly after discharge from the Medical Intensive Care Unit (MICU) and the potential effect of sleep quality in the MICU on those neurocognitive outcomes. The investigators hypothesize that post-ICU neurocognitive function and patient overall ICU sleep experience will improve through a pre-existing MICU sleep improvement initiative.

DETAILED DESCRIPTION:
Despite decades of scientific interest in evaluating sleep among critically ill patients, little is known about the effects of intensive care unit (ICU)-associated sleep disturbances on patient outcomes. Furthermore, few interventions have been rigorously evaluated to demonstrate efficacy in improving sleep in the ICU and associated patient outcomes. Post-ICU neurocognitive test performance data from this study will be linked to a pre-existing Quality Improvement (QI) project for patient sleep in the MICU. We hypothesize that patients' post-ICU neurocognitive performance (delirium status, attention, short-term memory, processing speed, and executive function) will positively correlate with scores from a previously-published Sleep in the Intensive Care Unit Questionnaire. In addition, we hypothesize that both neurocognitive performance and the Sleep in the Intensive Care Unit Questionnaire will improve during the multi-stage MICU-wide sleep QI project. Our project will provide valuable empirical evidence to help support guidelines for promoting sleep in the ICU setting.

ELIGIBILITY:
Inclusion Criteria:

* >=18 years old
* Spent at least one full night (i.e. 7pm to 7am) in the Johns Hopkins Hospital (JHH) Medical Intensive Care Unit (MICU).
* Discharged directly from MICU to an in-patient medical step-down or ward bed at JHH.

Exclusion Criteria:

* Previously enrolled in the study (i.e. repeat discharge from MICU)
* Pre-existing cognitive impairment, including hepatic encephalopathy, long-term alcohol abuse, and neurological disease (e.g., dementia, prior stroke, cerebral palsy, traumatic brain injury, active seizures)
* Unable to speak and/or understand English
* > 96 hours between MICU discharge and testing
* Visual or hearing impairment, inability to read, or inability to use a writing instrument preventing administration of the neurocognitive tests
* Spent at least one night in an ICU other than JHH MICU during current hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2010-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Digit span test score | within 96 hours of Intensive Care Unit (ICU) discharge

SECONDARY OUTCOMES:
Sleep in the ICU Questionnaire | within 96 hours of ICU discharge
Trail Making Test (Part A + B) times | within 96 hours of ICU discharge
Delirium status | within 96 hours of ICU discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States